CLINICAL TRIAL: NCT00254930
Title: Prospective Trial of Risperdal (Risperidone) Following Psychological Therapy for Challenging Behaviour in Learning Disabled Children
Brief Title: A Prospective Study of Risperdal (Risperidone) for the Treatment of Behavioral Disorder Following Psychological Therapy for Challenging Behavior in Learning Disabled Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005797
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2010-03

CONDITIONS: Learning Disorders; Child Behavior Disorders
Keywords: learning disorder; children; behaviour disorder; risperidone
MeSH Terms: conditions — Learning Disabilities; Child Behavior Disorders; Mental Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to assess whether risperidone (an antipsychotic medication) is safe and effective in treating behaviour disorder in learning disabled children, which does not improve with psychological therapy.

DETAILED DESCRIPTION:
There is a high incidence of behaviour disorder in people who are learning disabled. The purpose of this study is to assess whether risperidone is safe and effective in the treatment of learning disabled children diagnosed with behaviour disorder, which does not improve with psychological therapy. If the learning disability is very severe, or the behaviour disorder is very severe, such therapy is not appropriate and thus is not attempted; these patients are nevertheless eligible to participate in the study. At the beginning of treatment, the dose of risperidone is titrated, by gradual increase from 0.25 mg/day up to a maximum of 4 mg/day, based on therapeutic response, with decreases allowed in case of adverse reactions. Patients will be assessed over six months. The primary measure of effectiveness is the change compared to baseline in the total score on the Aberrant Behaviour Checklist (ABC). The EPSS is used to monitor the appearance of extrapyramidal symptoms. Based on results from other studies and the differences observed as a result of treatment, the investigator and his team expect to be able to detect a statistically and clinically significant result if data are available for 15 evaluable patients. Twenty patients will be recruited, taking account of possible drop outs. 0.25 mg of risperidone per day, taken orally, up to a maximum daily dose of 4 mg/day, for a treatment period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Axis II diagnosis of mental retardation
* behavioural and family therapy tried for 6 months but has failed
* in school, at least part time
* score of >=8 on hostility scale
* subject is otherwise healthy

Exclusion Criteria:

* Patients with a seizure disorder requiring repeated change of medication
* extrapyramidal symptoms not well controlled by medication
* abnormal and clinically significant electrocardiogram (ECG) changes
* history of tardive dyskinesia (a condition of uncontrollable movements of the tongue, lips, face, trunk, hands and feet that is seen in patients receiving long-term medication with certain types of antipsychotic drugs), or neuroleptic malignant syndrome (a rare condition in patients receiving antipsychotic medication in which patients may develop fever, sweating, unstable blood pressure, rigid muscles, and other symptoms, including changes in their normal mental state)
* known hypersensitivity to antipsychotic medications, including risperidone.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2003-09; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change compared to baseline in total score of the Aberrant Behaviour Checklist (ABC)

SECONDARY OUTCOMES:
Changes compared to baseline of Aberrant Behaviour Checklist (ABC) subclasses; hostility checklist; Clinical Global Impression (CGI) of severity; child quality of life rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.

REFERENCES:
- See also: Prospective trial of risperidone (Risperdal) following psychological therapy for challenging behaviour in learning disabled children — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=263&filename=CR005797_CSR.pdf